CLINICAL TRIAL: NCT00187005
Title: Total Therapy Study XIV for Newly Diagnosed Patients With Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Toxicity
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Ching-Hon Pui, MD / Principal Investigator, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOTXIV
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2008-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Prednisone; Dexamethasone; Vincristine; Daunorubicin; pegaspargase; Asparaginase; Methotrexate; Idarubicin; Etoposide; Cyclophosphamide; Cytarabine; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: Prednisone, Dexamethasone, Vincristine, Daunorubicin, PEG-L-asparaginase; Drug: L-asparaginase, Methotrexate, Idarubicin, Etoposide, Cyclophosphamide, Cytarabine, Mercaptopurine

INTERVENTIONS:
Drug: Prednisone, Dexamethasone, Vincristine, Daunorubicin, PEG-L-asparaginase — See Detailed Description section for details of treatment interventions.
Drug: L-asparaginase, Methotrexate, Idarubicin, Etoposide, Cyclophosphamide, Cytarabine, Mercaptopurine — See Detailed Description section for details of treatment interventions.

SUMMARY:
The main purpose of this study is to find out if radiation to the central nervous system (CNS) can be safely omitted with early intensification of chemotherapy and chemotherapy given directly to the CNS. Another purpose is to find out if survival of children with ALL can be improved with risk-directed therapy given on this protocol.

DETAILED DESCRIPTION:
There are multiple secondary objectives in this trial:

* To estimate the overall event-free survival of patients treated with risk-directed therapy
* To identify the plasma methotrexate (MTX) concentrations that produce maximum intracellular accumulation of active metabolites (methotrexate polyglutamates, MTXPG) in vivo, in relation to major cell lineage and genotype
* To determine the relation between MTXPG accumulation in leukemic lymphoblasts and antileukemic effects, as measured by the inhibition of de novo purine synthesis, and by the decrease in circulating blasts during the 4 days after initiation of single-agent high-dose methotrexate treatment
* To determine if plasma MTX concentrations exceeding those required for maximum MTXPG accumulation cause a paradoxical decrease in the accumulation of long-chain MTXPG in lymphoblasts, (e.g., due to "feedback inhibition" of folypolyglutamate synthetase)
* To determine if there are significant differences in lymphoblast uptake of MTX and expression of the reduced folate carrier in T-lineage vs B-lineage lymphoblasts, and in hyperdiploid vs non-hyperdiploid B-lineage lymphoblasts
* To investigate whether atovaquone (ATQ) is as effective as trimethoprim-sulfamethoxazole (TMP-SMZ) in preventing Pneumocystis carinii pneumonitis (PCP)
* To investigate whether or not the administration of G-CSF at the onset of febrile episodes in neutropenia patients after induction or any of the two reinductions will affect the extent and duration of fever.
* To determine whether levels of minimal residual disease in peripheral blood (PB) reflect those measured in the bone marrow (BM) by immunologic or molecular techniques
* To assess the degree of DNA damage in somatic cells (leukocytes) during treatment
* To explore whether genetic polymorphisms of enzymes important in metabolism of antileukemic agents (e.g. methylene tetrahydrofolate reductase, thiopurine methyltransferase, glutathione transferases) are correlated with MTX pharmacology in lymphoblasts, acute toxicities and long-term outcome
* To explore whether the development of anti-asparaginase antibodies or CSF depletion of asparaginase is correlated with acute toxicities and long-term outcome
* To assess the relation between MRI changes of brain (especially white matter abnormalities) from HDMTX and intrathecal treatment, neurologic and cognitive deficits, CSF levels of homocysteines and diminished quality of life
* To investigate whether early MRI changes are related to late MRI abnormalities, neurologic and cognitive deficits, and diminished quality of life
* To correlate changes in MRI, neurologic or cognitive deficits and diminished quality of life with selected pharmacokinetic variables
* To determine the prevalence of low bone density and to correlate this complication with potential risk factors

Details of Treatment Interventions:

Treatment will consist of three main phases, Remission Induction (including an Upfront HDMTX Window), Consolidation, and Continuation.

Window Therapy Upfront HDMTX is considered the first part of remission induction treatment. HDMTX will be given by vein over 24 hours (one day). MTX 500 mg/m2 for standard risk and 250 mg/m2 for low-risk cases will be given over 1 hour, followed immediately by maintenance infusion (4500 mg/m2 for standard/high-risk or 2250 mg/m2 for low-risk cases) over 23 hours.

Remission Induction Therapy (6-7 weeks) The remaining induction treatment will begin with Prednisone 40 mg/m2/day PO (tid) Days 5-32, Vincristine 1.5 mg/m2/week IV days 5, 12, 19, 26, Daunorubicin 25 mg/m2/week IV days 5, 12, L-asparaginase 10,000 U/m2/dose IM (thrice weekly) days 6, 8, 10, 12, 14, 16 (19, 21, 23), and triple intrathecal treatment, followed by Etoposide 300 mg/m2/dose IV over 2 hr days 26, 29, 33, plus Cytarabine 300 mg/m2/dose IV over 2 hr Days 26, 29, 33.

Triple intrathecal chemotherapy (MHA) is used for the remaining treatment with dosages based on age Frequency and total number of triple intrathecal treatment for Remission Induction are based on the patient's risk of CNS relapse.

Consolidation (2 weeks) Patients receive High dose Methotrexate (HDMTX) 2.5 gm/m2 (low-risk) or 5 gm/m2 (standard-or-high-risk) IV over 24 hr days 1 and 8 and 6-Mercaptopurine 25 mg/m2/day PO days 1 to 14. All patients will receive triple intrathecal therapy weekly for two doses on Days 1 and 8.

Continuation treatment (120 weeks for girls and 146 weeks for boys) Post-remission continuation treatment begins 7 days after the second course of HDMTX of the consolidation treatment, provided that the ANC ≥300/mm3 and platelet count ≥ 50 x 109/L. Continuation treatment will be 120 weeks for girls and 146 weeks for boys and differs according to the risk classification.

Reinduction Treatment This phase of treatment will be started at weeks 12 and 28 after bone marrow examination confirms complete remission.

Reinduction treatment will be given twice:

Weeks 12 to 16 and week 28 to 32 for standard/high risk cases; weeks 12 to 15 and weeks 28-31 for low-risk cases. Leucovorin rescue (5 mg/m2) will be given at 24 and 30 hours after the intrathecal treatment during both remission reinduction treatments. No chemotherapy will be given weeks 16 and 32 for standard/high risk patients.

Standard- or High-Risk Leukemia

* DEX (dexamethasone) 8 mg/m2 PO daily (tid) x 7 days and VCR (vincristine) 1.5 mg/m2 IV push (max. 2 mg) will be given weeks 1, 5, 9, 17, 21, 25, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, 81, 85, 89, 93, 97, 101, 105, 109, 113, and 117.
* VP16 (etoposide) 300 mg/m2 IV over 2 hours and CTX (cyclophosphamide) 300 mg/m2 IV short infusion will be given weeks 2, 6, 10, 18, 22, 26, 34, 38, 42, 46, 50, 54, 58, 62, 66, 70, 74, 78, 82, 86, 90, and 94.
* 6MP (6-mercaptopurine) 75 mg/m2 PO daily x 7 days and MTX (methotrexate) 40 mg/m2 IV or IM weeks 3, 8, 11, 19, 24, 27, 35, 39, 40, 43, 47, 48, 51, 55, 56, 59, 63, 64, 67, 71, 72, 75, 79, 80, 83, 87, 88, 91, 95, 96, 98, 99, 102, 103, 104, 106, 107, 110, 111, 112, 114, 115, 118, 119, and 120, and weeks 121-146 for boys.
* MTX (methotrexate) 40 mg/m2 IV or IM and Ara-C (cytarabine) 300 mg/m2 IV push will be given weeks4, 20, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, and 116.
* 6MP (6-mercaptopurine) 75 mg/m2 PO daily x 7 days and HDMTX 5 gm/ gm/m2 will be given week 7 and 23.
* HDMTX 5 gm/ gm/m2 and Ara-C (cytarabine) 300 mg/m2 IV push will be given weeks 15 and 31.

Reinduction Treatment-Standard/High Risk

* DEX (dexamethasone) 8 mg/m2 PO daily (tid) days 1-21,
* VCR (vincristine) 1.5 mg/m2/week IV (max. 2 mg) days 1, 8, and 15
* PEG-asparaginase 2500 U/m2/week IM weeks 28-31, days 8, and 15
* Idarubicin 5 mg/m2/week IV days 1 and 8
* HDMTX 5 gm/m2 IV day 22
* ITMHA (methotrexate+hydrocortisone+ara-C), age dependent, IT day 1
* High-dose cytarabine 2 gm/m2 IV q 12 hr Days 23, and 24 Low Risk
* 6MP (6-mercaptopurine) 75 mg/m2 PO daily x 7 days and MTX (methotrexate) 40 mg/m2 IV or IM weeks 1, 2, 3, 4, 6, 8, 10,, 11, 16, 18- 20, 22, 24, 26, 27, 32, 34- 36, 38-40, 42- 44, 46-48, 50-52, 54-56, 58-60, 62-64, 66-68, 70-72, 74-76, 78-80, 82-84, 86-88, 90-92, 94-96, 98-100, 102-104, 106-108, 110-112, 114-116, 118-120 and weeks 121-146 for boys.
* 6MP (6-mercaptopurine) 75 mg/m2 PO daily x 7 days, MTX (methotrexate) 40 mg/m2 IV or IM, DEX (dexamethasone) 8 mg/m2 PO daily (tid) x 7 days and VCR (vincristine) 1.5 mg/m2 IV push (max. 2 mg) weeks 5, 9, 17, 21, 25, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, 81, 85, 89, 93, 97, 101, 105, 109, 113, and 117.
* 6MP (6-mercaptopurine) 75 mg/m2 PO daily x 7 days and HDMTX 2.5 gm/m2 weeks 7, 15, 23 and 31.

Reinduction Treatment-Low Risk

* DEX (dexamethasone) 8 mg/m2 PO daily days 1-21,
* VCR (vincristine) 1.5 mg/m2/week IV push (max. 2 mg) days 1, 8, and 15
* PEG-asparaginase 2500 U/m2/week IM days 8, and 15
* Idarubicin 5 mg/m2/week IV day 1
* HDMTX 2.5 gm/m2 day 22
* ITMHA (methotrexate+hydrocortisone+ara-C), age dependent, IT day 1 and 22
* 6 MP 75 mg/m2/day PO days 22-28 IT Chemotherapy
* Triple intrathecal treatment will be given to low-risk cases with CNS-1 status on weeks 1, 2, 7, 12, 15, 23, 28, 31, 39, 47, and 54.
* Triple intrathecal treatment will be given to low-risk cases with CNS-2 or traumatic CSF status on weeks 1, 2, 7, 12, 15, 19, 23, 28, 31, 36, 39, 43, 47, and 54.
* Triple intrathecal treatment will be given to standard/high-risk cases on weeks 1, 2, 7, 12, 19, 23, 28, 36, 39, 43, 47, and 54.
* Triple intrathecal treatment will be given to other standard/high-risk cases with WBC ≥100 x 109/L, T-cell ALL with WBC ≥50 x 109/L, presence of Philadelphia chromosome, MLL rearrangement, near haploidy, or CNS-3 status on weeks 1, 2, 7, 12, 19, 23, 28, 36, 39, 43, 47, 54, 64, 72, 80, and 88.

Hematopoietic Stem Cell Transplantation Patients who meet the criteria of high-risk ALL will be offered the option of transplantation with a matched, related or unrelated donor. However, if the option is declined or if a suitable donor is not available, the patient will remain on study and continue to receive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-B-cell leukemia by immunophenotyping (e.g. T-cell, B-cell precursor, or acute undifferentiated leukemia)
* Ages less than or equal to 18 years of age
* One week or less of prior therapy, limited to glucocorticoids, vinca alkaloids, emergency radiation therapy to the mediastinum and one dose of intrathecal chemotherapy Exclusion Criteria
* Participants greater than 18 years of age

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 1998-07; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
To determine if CNS irradiation can be safely omitted with early intensification of systemic and intrathecal chemotherapy. | Unable to determine

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hon Pui, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St.Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Hammond TG, Hu A, Hammond JM, Relling MV, Underwood JL. Detection of point mutations on a DNA microchip Clinical Immunology Newsletter 19(12):121-6, 1999.
- [Background] Pui CH, Mahmoud HH, Wiley JM, Woods GM, Leverger G, Camitta B, Hastings C, Blaney SM, Relling MV, Reaman GH. Recombinant urate oxidase for the prophylaxis or treatment of hyperuricemia in patients With leukemia or lymphoma. J Clin Oncol. 2001 Feb 1;19(3):697-704. doi: 10.1200/JCO.2001.19.3.697. PMID 11157020
- [Background] Pui CH, Jeha S, Irwin D, Camitta B. Recombinant urate oxidase (rasburicase) in the prevention and treatment of malignancy-associated hyperuricemia in pediatric and adult patients: results of a compassionate-use trial. Leukemia. 2001 Oct;15(10):1505-9. doi: 10.1038/sj.leu.2402235. PMID 11587206
- [Background] Panetta JC, Yanishevski Y, Pui CH, Sandlund JT, Rubnitz J, Rivera GK, Ribeiro R, Evans WE, Relling MV. A mathematical model of in vivo methotrexate accumulation in acute lymphoblastic leukemia. Cancer Chemother Pharmacol. 2002 Nov;50(5):419-28. doi: 10.1007/s00280-002-0511-x. Epub 2002 Sep 24. PMID 12439601
- [Background] Coustan-Smith E, Sancho J, Behm FG, Hancock ML, Razzouk BI, Ribeiro RC, Rivera GK, Rubnitz JE, Sandlund JT, Pui CH, Campana D. Prognostic importance of measuring early clearance of leukemic cells by flow cytometry in childhood acute lymphoblastic leukemia. Blood. 2002 Jul 1;100(1):52-8. doi: 10.1182/blood-2002-01-0006. PMID 12070008
- [Background] Coustan-Smith E, Sancho J, Hancock ML, Razzouk BI, Ribeiro RC, Rivera GK, Rubnitz JE, Sandlund JT, Pui CH, Campana D. Use of peripheral blood instead of bone marrow to monitor residual disease in children with acute lymphoblastic leukemia. Blood. 2002 Oct 1;100(7):2399-402. doi: 10.1182/blood-2002-04-1130. PMID 12239148
- [Background] Yeoh EJ, Ross ME, Shurtleff SA, Williams WK, Patel D, Mahfouz R, Behm FG, Raimondi SC, Relling MV, Patel A, Cheng C, Campana D, Wilkins D, Zhou X, Li J, Liu H, Pui CH, Evans WE, Naeve C, Wong L, Downing JR. Classification, subtype discovery, and prediction of outcome in pediatric acute lymphoblastic leukemia by gene expression profiling. Cancer Cell. 2002 Mar;1(2):133-43. doi: 10.1016/s1535-6108(02)00032-6. PMID 12086872
- [Background] Panetta JC, Wall A, Pui CH, Relling MV, Evans WE. Methotrexate intracellular disposition in acute lymphoblastic leukemia: a mathematical model of gamma-glutamyl hydrolase activity. Clin Cancer Res. 2002 Jul;8(7):2423-9. PMID 12114448
- [Background] Cheok MH, Yang W, Pui CH, Downing JR, Cheng C, Naeve CW, Relling MV, Evans WE. Treatment-specific changes in gene expression discriminate in vivo drug response in human leukemia cells. Nat Genet. 2003 May;34(1):85-90. doi: 10.1038/ng1151. PMID 12704389
- [Background] Kishi S, Griener J, Cheng C, Das S, Cook EH, Pei D, Hudson M, Rubnitz J, Sandlund JT, Pui CH, Relling MV. Homocysteine, pharmacogenetics, and neurotoxicity in children with leukemia. J Clin Oncol. 2003 Aug 15;21(16):3084-91. doi: 10.1200/JCO.2003.07.056. PMID 12915598
- [Background] Hinds PS, Gattuso JS, Fletcher A, Baker E, Coleman B, Jackson T, Jacobs-Levine A, June D, Rai SN, Lensing S, Pui CH. Quality of life as conveyed by pediatric patients with cancer. Qual Life Res. 2004 May;13(4):761-72. doi: 10.1023/B:QURE.0000021697.43165.87. PMID 15129886
- [Background] Hak LJ, Relling MV, Cheng C, Pei D, Wang B, Sandlund JT, Rubnitz J, Pui CH. Asparaginase pharmacodynamics differ by formulation among children with newly diagnosed acute lymphoblastic leukemia. Leukemia. 2004 Jun;18(6):1072-7. doi: 10.1038/sj.leu.2403351. PMID 15057247
- [Background] Neale GA, Coustan-Smith E, Stow P, Pan Q, Chen X, Pui CH, Campana D. Comparative analysis of flow cytometry and polymerase chain reaction for the detection of minimal residual disease in childhood acute lymphoblastic leukemia. Leukemia. 2004 May;18(5):934-8. doi: 10.1038/sj.leu.2403348. PMID 15029212
- [Background] Cheng Q, Wu B, Kager L, Panetta JC, Zheng J, Pui CH, Relling MV, Evans WE. A substrate specific functional polymorphism of human gamma-glutamyl hydrolase alters catalytic activity and methotrexate polyglutamate accumulation in acute lymphoblastic leukaemia cells. Pharmacogenetics. 2004 Aug;14(8):557-67. doi: 10.1097/01.fpc.0000114761.78957.7e. PMID 15284538
- [Background] Rubnitz JE, Lensing S, Zhou Y, Sandlund JT, Razzouk BI, Ribeiro RC, Pui CH. Death during induction therapy and first remission of acute leukemia in childhood: the St. Jude experience. Cancer. 2004 Oct 1;101(7):1677-84. doi: 10.1002/cncr.20532. PMID 15378506
- [Background] Glass JO, Reddick WE, Reeves C, Pui CH. Improving the segmentation of therapy-induced leukoencephalopathy in children with acute lymphoblastic leukemia using a priori information and a gradient magnitude threshold. Magn Reson Med. 2004 Dec;52(6):1336-41. doi: 10.1002/mrm.20259. PMID 15562471
- [Background] Cox CL, Lensing S, Rai SN, Hinds P, Burghen E, Pui CH. Proxy assessment of quality of life in pediatric clinical trials: application of the Health Utilities Index 3. Qual Life Res. 2005 May;14(4):1045-56. doi: 10.1007/s11136-004-4714-y. PMID 16041900
- [Background] Reddick WE, Glass JO, Helton KJ, Langston JW, Xiong X, Wu S, Pui CH. Prevalence of leukoencephalopathy in children treated for acute lymphoblastic leukemia with high-dose methotrexate. AJNR Am J Neuroradiol. 2005 May;26(5):1263-9. PMID 15891195
- [Background] Lowe EJ, Pui CH, Hancock ML, Geiger TL, Khan RB, Sandlund JT. Early complications in children with acute lymphoblastic leukemia presenting with hyperleukocytosis. Pediatr Blood Cancer. 2005 Jul;45(1):10-5. doi: 10.1002/pbc.20178. PMID 15547931
- [Background] Cheng Q, Yang W, Raimondi SC, Pui CH, Relling MV, Evans WE. Karyotypic abnormalities create discordance of germline genotype and cancer cell phenotypes. Nat Genet. 2005 Aug;37(8):878-82. doi: 10.1038/ng1612. Epub 2005 Jul 24. PMID 16041371
- [Background] Zaza G, Cheok M, Yang W, Panetta JC, Pui CH, Relling MV, Evans WE. Gene expression and thioguanine nucleotide disposition in acute lymphoblastic leukemia after in vivo mercaptopurine treatment. Blood. 2005 Sep 1;106(5):1778-85. doi: 10.1182/blood-2005-01-0143. Epub 2005 May 19. PMID 15905191
- [Background] Pui CH, Pei D, Sandlund JT, Campana D, Ribeiro RC, Razzouk BI, Rubnitz JE, Howard SC, Hijiya N, Jeha S, Cheng C, Downing JR, Evans WE, Relling MV, Hudson M. Risk of adverse events after completion of therapy for childhood acute lymphoblastic leukemia. J Clin Oncol. 2005 Nov 1;23(31):7936-41. doi: 10.1200/JCO.2004.01.0033. PMID 16258093
- [Background] Pui CH, Evans WE. Treatment of acute lymphoblastic leukemia. N Engl J Med. 2006 Jan 12;354(2):166-78. doi: 10.1056/NEJMra052603. No abstract available. PMID 16407512
- [Background] Flotho C, Coustan-Smith E, Pei D, Iwamoto S, Song G, Cheng C, Pui CH, Downing JR, Campana D. Genes contributing to minimal residual disease in childhood acute lymphoblastic leukemia: prognostic significance of CASP8AP2. Blood. 2006 Aug 1;108(3):1050-7. doi: 10.1182/blood-2006-01-0322. Epub 2006 Apr 20. PMID 16627760
- [Background] Raimondi SC, Zhou Y, Shurtleff SA, Rubnitz JE, Pui CH, Behm FG. Near-triploidy and near-tetraploidy in childhood acute lymphoblastic leukemia: association with B-lineage blast cells carrying the ETV6-RUNX1 fusion, T-lineage immunophenotype, and favorable outcome. Cancer Genet Cytogenet. 2006 Aug;169(1):50-7. doi: 10.1016/j.cancergencyto.2006.04.006. PMID 16875937
- [Background] Jeha S, Behm F, Pei D, Sandlund JT, Ribeiro RC, Razzouk BI, Rubnitz JE, Hijiya N, Howard SC, Cheng C, Pui CH. Prognostic significance of CD20 expression in childhood B-cell precursor acute lymphoblastic leukemia. Blood. 2006 Nov 15;108(10):3302-4. doi: 10.1182/blood-2006-04-016709. Epub 2006 Aug 8. PMID 16896151
- [Background] Hijiya N, Panetta JC, Zhou Y, Kyzer EP, Howard SC, Jeha S, Razzouk BI, Ribeiro RC, Rubnitz JE, Hudson MM, Sandlund JT, Pui CH, Relling MV. Body mass index does not influence pharmacokinetics or outcome of treatment in children with acute lymphoblastic leukemia. Blood. 2006 Dec 15;108(13):3997-4002. doi: 10.1182/blood-2006-05-024414. Epub 2006 Aug 17. PMID 16917005
- [Background] Madden RM, Pui CH, Hughes WT, Flynn PM, Leung W. Prophylaxis of Pneumocystis carinii pneumonia with atovaquone in children with leukemia. Cancer. 2007 Apr 15;109(8):1654-8. doi: 10.1002/cncr.22562. PMID 17345613
- [Background] Relling MV, Yang W, Das S, Cook EH, Rosner GL, Neel M, Howard S, Ribeiro R, Sandlund JT, Pui CH, Kaste SC. Pharmacogenetic risk factors for osteonecrosis of the hip among children with leukemia. J Clin Oncol. 2004 Oct 1;22(19):3930-6. doi: 10.1200/JCO.2004.11.020. PMID 15459215
- [Background] Reddick WE, Glass JO, Helton KJ, Langston JW, Li CS, Pui CH. A quantitative MR imaging assessment of leukoencephalopathy in children treated for acute lymphoblastic leukemia without irradiation. AJNR Am J Neuroradiol. 2005 Oct;26(9):2371-7. PMID 16219848
- [Background] Coustan-Smith E, Ribeiro RC, Stow P, Zhou Y, Pui CH, Rivera GK, Pedrosa F, Campana D. A simplified flow cytometric assay identifies children with acute lymphoblastic leukemia who have a superior clinical outcome. Blood. 2006 Jul 1;108(1):97-102. doi: 10.1182/blood-2006-01-0066. Epub 2006 Mar 14. PMID 16537802
- See also: St. Jude Children's Research Hospital — http://www.stjude.org